CLINICAL TRIAL: NCT06292416
Title: Effects of Mirror Therapy With Sensory Motor Training on Upper Limb Functions and Quality of Movement in Children With Hemiplegic Cerebral Palsy
Brief Title: Mirror Therapy With Sensory Motor Training in Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0257Huma Saleem
Record Dates: First submitted 2023-12-26; First posted 2024-03-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Hemiplegic; Mirror Therapy; Strength training
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be kept blind about the intervention which the patients will be receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy with sensory motor training. (Experimental): 1. Visual perception activities
  2. Body awareness
  3. Tactile perception.
  4. Visual-motor coordination training
  The child will be seated on a chair and a 30*30 cm mirror will set up on a table in front of them. The affected hand will be placed behind the mirror so that the image of a healthy hand can be seen clearly
  Interventions: Other: Experimental: Mirror therapy with sensory motor training.
- Mirror Therapy with motor training. (Experimental): supination-pronation, wrist flexion-extension, finger flexion-extension, abduction, adduction, opposition
  Interventions: Other: Experimental: Mirror Therapy with motor training
- Motor Training (Other): 1. Holding objects
  2. Stabilize objects
  3. manipulate objects
  Interventions: Other: Experimental: Motor Training

INTERVENTIONS:
Other: Experimental: Mirror therapy with sensory motor training. — Block design, finding shapes in pictures, puzzles, matching geometric shapes and letters, numbers, and classification.
  Pointing to the body parts, life-size drawing, turning left and right side and awareness of the body parts through touch.
  feeling various textures, touching boards, and feeling shapes. Ocular-pursuit training, moving ball and pegboard activities During the sessions, subjects were asked to try and do the same movement with the paretic hand simultaneously The patients will be asked to repeat each movement 20 times per set for three sets, with a 2-minute break between sets.
  Session will last for 45 mins
  Arms: Mirror therapy with sensory motor training.
Other: Experimental: Mirror Therapy with motor training — the participant is asked to perform a forearm movement sting on the paretic side while the subjects look into the mirror, watching the image of their non-involved hand and thus seeing the reflection of the hand movement projected over the involved hand. During the sessions subjects were asked to try and do the same movement with the paretic hand simultaneously. movement was repeated 20 times per set for three sets, with a 2-minute break between sets
  Arms: Mirror Therapy with motor training.
Other: Experimental: Motor Training — 1. Holding object with two hands, clapping, banging objects together.
  2. Stabilize objects with one hand while the other is manipulating (holding paper while coloring, holding a container while putting objects in)
  3. manipulate objects with both hands simultaneously (stringing beads, tying a knot),
  4. ask child to padlock in which a key can be put into, markers with caps to put on, a box with a lid and objects to put inside the box
  5. hold a cup with one hand while putting object in with other hand
  6. Buttoning with both hands, tying a bow. doing craft project, fitting blocks together
  Arms: Motor Training

SUMMARY:
The study compares two interventions in CP children: mirror therapy with sensory motor training versus mirror therapy with motor training. Mirror therapy works by manipulating the brain out of pain, ultimately improving movement in patients with one-sided paralysis. It can be used in combination with other therapies to assist patients with cerebral palsy in retraining the brains, restoring function, and enhancing the overall quality of life. The purpose of this study is to use a combination of Mirror therapy with sensory motor training and motor training and observe which one of these combinations has the most desirable effects in improving movement and quality of life in CP Children

DETAILED DESCRIPTION:
The neurodevelopmental disorder known as cerebral palsy (CP) is caused by damage to the developing brain and is characterized by abnormalities of muscle tone, mobility, and motor skills. A person with cerebral palsy can be classified according to how it affects movement, the area of the body that is affected, and how severe the effects are. Children with hemiplegic cerebral palsy have a variety of motor and sensory deficits in the upper limb, which makes it more difficult to perform everyday tasks including reaching, gripping, releasing, and manipulating things. The movement produced by constraints on the less-affected hand and extensive training on the more-affected hand aims to enhance upper limb function in hemiparetic youngsters. One such intervention to improve the motor function of these patients is the use of mirror therapy. Mirror therapy is one of the more recent approaches to helping the more severely afflicted upper extremities regain function after stroke. During mirror therapy, a mirror is held in the patient's midsagittal plane, reflecting the less-affected side as though it were the more-affected side. In this arrangement, the motions of the less affected extremity give the impression that the more affected extremity is moving normally. Mirror treatment is easy to use, reasonably priced, and non-intrusive. This makes it a promising and secure complement to hemiparesis therapy for children. Sensorimotor training involves proprioceptive and balance exercises that were developed to help individuals suffering from chronic musculoskeletal pain syndromes. Repetitive sensorimotor training may increase the responsiveness of nociceptive-evoked potentials. Motor training, on the other hand, focuses on skill acquisition through repetition. Through this study, the investigator wants to use a combination of techniques to improve upper limb function and quality of movement in patients with CP

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 12 years
* Lack of use of the affected upper limb
* Level I-III of the Manual Ability Classification System (MACS)
* Level I-III in the Gross Motor Function Classification System (GMFCS)

Exclusion Criteria:

* Disease not associated with congenital hemiplegia
* Presence of contractures in the affected upper limb affecting the functional movement
* Surgery in the six months previously to the treatment
* Botulinum toxin in the two months previously to or during the intervention
* Pharmacologically uncontrolled epilepsy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
The Melbourne Assessment of Unilateral Upper Limb Function (Melbourne Assessment) | Assessment will be done at 6th week by outcome measuring tool
  It is an evaluation tool that objectively measures upper-extremity function in children with cerebral palsy. The total score is 122, which is the maximum, whereas the minimum score is 0. It is Reported as a percentage, with higher scores reflecting greater quality of upper-limb movement
Jebsen Taylor Hand dysfunction test | 6 weeks
  It measures the fine and gross motor function of the hands. The results are measured by timing the time taken to accomplish each task.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Saleem, MS NMPT*, Principal Investigator — Riphah International Univerisity; Ammara Abbas, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Eliya care Centre Faisalabad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No